CLINICAL TRIAL: NCT03236532
Title: Impact of Physical Exercise Associated With Glutamine Supplementation in Health Indicators of People Living With HIV/AIDS
Brief Title: Effect of Supplementation With Glutamine and Exercise in Women With HIV/AIDS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: State University of Maringá (Other)
Collaborators: Conselho Nacional de Desenvolvimento Científico e Tecnológico (Other Government)
Responsible Party: Principal Investigator, Ademar Avelar de Almeida Junior, Principal Investigator, State University of Maringá
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: State University of Maringá
Record Dates: First submitted 2017-07-28; First posted 2017-08-02 (Actual); Last update posted 2017-08-22 (Actual); Status verified 2017-08

CONDITIONS: Glutamine; Metabolic Disorder; Physical Activity
Keywords: HIV/AIDS; Resistance training, supplementation
MeSH Terms: conditions — Metabolic Diseases; Motor Activity; Acquired Immunodeficiency Syndrome | interventions — Glutamine; Exercise; maltodextrin

STUDY DESIGN:
Intervention Model Description: In the first stage, the participants were initially randomly separated in a double-blind way in order to ingest either the GDP (Condition 1) or maltodextrin as a placebo (Condition 2) for seven days. On the seventh and last day of supplementation, they were submitted to the resistance training session. Before and immediately after the exercise session, the cognitive tests were applied. After these procedures there was a one-week rest period (step 2). Then the procedures performed in the first step were repeated (step 3). However, the group that had received GDP started to receive maltodextrin, and the group who had received maltodextrin started to receive GDP, adopting, thus, a randomized double-blind crossover design.
Who Masked: Participant, Investigator
Masking Description: The substances were packed in sachets containing GDP (glutamine) or maltodextrin (placebo). The packages were identical and the substances used had a similar color and texture. An external subject organized group division and substances delivery.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Glutamine and exercise (Experimental): Glutamine dipeptide (20g/day) in 300 ml of water and ingest it after lunch during 7 days. In case of forgetfulness, they were suggested to ingest it soon after dinner. All participants were instructed to maintain their routine eating habits throughout the duration of the study. On the seventh and last day of supplementation, they were submitted to the resistance training session.
  Interventions: Dietary Supplement: Glutamine and exercise
- Maltodextrin and exercise (Placebo Comparator): Maltodextrin (20g/day) in 300 ml of water and ingest it after lunch during 7 days. In case of forgetfulness, they were suggested to ingest it soon after dinner. All participants were instructed to maintain their routine eating habits throughout the duration of the study. On the seventh and last day of supplementation, they were submitted to the resistance training session.
  Interventions: Dietary Supplement: Maltodextrin and exercise

INTERVENTIONS:
Dietary Supplement: Glutamine and exercise
  Arms: Glutamine and exercise
Dietary Supplement: Maltodextrin and exercise
  Arms: Maltodextrin and exercise

SUMMARY:
This study aimed to investigate the effect of an exercise session with weights associated with glutamine dipeptide (GLD) supplementation on cognitive function of people living with HIV/ AIDS. The sample consisted of 10 HIV+ women, who used the Antiretroviral Therapy Highly Active. The participants were randomized in a double-blind procedure to receive seven days of supplementation GLD or placebo (PLA). At the end of this first period, the participants held a workout with weights with cognitive assessments before and immediately after the session. To evaluate oxidative stress markers blood samples were collected before and 1 hour and 2 hours after the session.Then the participants rested for 7 days for the initial stocks of glutamine return to baseline levels (washout). Following was realized the crossing of the groups, so those who had received the GLD in the first week spent extra for 7 days with PLA and vice versa, and then they repeated evaluations and exercise session. The exercise session consisted of seven resistance exercises involving different muscle groups, with three sets of 8-12 repetitions with an interval of 90 seconds between sets and 120 seconds between the exercises. Stroop test was used to cognitive assessments, which aims to assess selective attention and inhibitory control over the color of conflict and word, and the N-back test, responsible for evaluating the central executive component of working memory by stimuli visual. Oxidative stress markers (TBARS, FOX, GSH, GSSG, AOPP) were analyzed in plasma samples.

DETAILED DESCRIPTION:
The aim of the present study was to investigate the effect of a short period of supplementation with glutamine dipeptide (GDP) in the acute responses to resistance training on people living with HIV/AIDS i the following healthy indicators: executive functions, stress oxidative markers, cardiovascular functions, inflammatory markers and biochemical markers.

Participants 14 women diagnosed with HIV+ participated in this study. As inclusion criteria, they should be over 18 years old; they should have regularly been using the Antiretroviral Therapy (ART) for more than six months; they should have a stabilized clinical picture and viral load; they should not have participated in physical training programs during the preceding six months; they should not show acute or chronic inflammations that could affect the practice of physical exercise; they should not have psychiatric disorders; and they should not be pregnant.

The individuals who met the inclusion criteria received clinical evaluation by the infectious physician responsible for the treatment based on the history of each patient, the laboratory tests and the clinical picture.

The study was approved by the Standing Committee on Ethical Research with Humans of the State University of Maringá - PR - Brazil. The volunteers signed the Free Informed Consent Form, after being informed about the study proposal and the procedures they would be submitted to.

During the study period, four participants were not able to attend all the evaluations and were excluded from the final analysis. Therefore, 10 women participated in all the procedures and were part of the final sample of the study.

Experimental design The study had a total duration of five weeks divided into two phases. The first phase lasted two weeks and was characterized by the familiarization with the exercises that would be done in the second phase. This protocol consisted of four sessions of exercises, every 48 hours, which submitted the individuals to the same procedures that would be done in the second phase. Four familiarization sessions were chosen, one of which was aimed at learning the exercises without the insertion of loads. Then, the participants could rest for a week before starting the second phase.

The second phase consisted of three stages; each of them lasted one week. In the first stage, the participants were initially randomly separated in a double-blind way in order to ingest either the GDP (Condition 1) or maltodextrin as a placebo (Condition 2) for seven days. On the seventh and last day of supplementation, they were submitted to the resistance training session. Before the exercise session the cognitive tests were applied, blood samples were collected for analysis of biochemical, inflammatory and oxidative stress markers. Immediately after the exercise session the cognitive tests were repeated. Blood samples were also collected 1 and 2 hours after the exercise training. Cardiovascular functions were monitorated during 1 hour after the exercise session, every 10 minutes. After these procedures there was one-week rest period (step 2). Then, the procedures performed in the first step were repeated (step 3). However, the group that had received GDP started to receive maltodextrin, and the group who had received maltodextrin started to receive GDP, adopting, thus, a randomized double-blind crossover design.

The resistance training protocol The exercises were based on the Guideline for the prescription of exercise to be given to people with HIV/AIDS. The training session consisted of seven exercises with weights (chest press, leg press 45º, lat pulldown machine, knee extension, triceps pulley, knee curl, Scott biceps curl machine) involving different muscle groups with three series per exercise.

The recovery interval adopted was of 90 seconds between the series and 120 seconds between exercises. The number of repetitions used in each one of these series was of 8-12 repetitions by applying the method of fixed loads. The loads were compatible with the number of repetitions stipulated for each exercise. The load determination occurred during familiarization sessions.

The OMNI Resistance Exercise Scale (OMNI-RES) of effort subjective perception was used to determine and control the loads of each exercise. The loads used during the experimental sessions corresponded to the intensity equivalent to the interval from five to seven (5-7) of the OMNI-RES scale.

In order to achieve such a purpose, prior to the beginning of familiarization with the exercises, the OMNI-RES scale anchoring was performed. This procedure consists of placing the patient in the smallest and highest possible load in each exercise so that he/she can differentiate a smaller and a greater subjective perception of effort.

Supplementation Protocol The participants were randomly double-blinded indicated to receive either GDP (20g/day) or maltodextrin (20g/day) according to the literature. The substances were packed in sachets containing GDP or maltodextrin (placebo). The packages were identical and the substances used had a similar color and texture. Participants were instructed to dilute GDP or maltodextrin in 300 ml of water and ingest it after lunch. In case of forgetfulness, they were suggested to ingest it soon after dinner. All participants were instructed to maintain their routine eating habits throughout the duration of the study.

Evaluation of the cognitive status Considering the general evaluation of possible cognitive impairments, the Mini Mental State Examination (MMSE) was used, which provides information on different cognitive parameters, considering the level of education of the individual evaluated.

In order to assess the indicatives of HIV-associated dementia the International HIV Dementia Scale was applied.

Executive Functions The Victoria Stroop color-word test was used to evaluate the executive functions, which consists of 72 stimuli, distributed in three cards with 24 items each (A, B, C). The subject must verbalize the name of the colors with which the stimuli of each card were printed as quickly as possible; the time spent to read each of the cards separately was registered. The latency time, which is determined by the difference between the time spent with the responses to the three cards, was used to evaluate selective attention and inhibitory control.

The n-back test was used to evaluate the operational memory. Visual stimuli were used in this study, which were represented by colors, divided into three levels (N1, N2, and N3) with 150 stimuli each. The score of each participant was obtained from the percentage values of the hits recorded in the three levels in a computerized version of the test.

Biochemical analysis Blood samples (10ml) were collected by venose puncture in heparinized vacutainer® tubes. Plasma glucose concentration were determined both using a glucose analyzer and using standard kit. Total cholesterol, HDL cholesterol and triglycerides were analysed by standard methods.

Inflammatory markers Plasma samples were also used to analyse interleukins 2, 6, 8 and 10 and TNFα using standard kits.

Oxidative stress markers Plasma malondialdehyde (MDA) was determined by high-performance liquid chromatography (UV/VIS SPD-20A SHIMADZU, Kioto, Japan) as described by Nielsen et al. Thiobarbituric acid reactive substances (TBARS) and Total hydroperoxide (FOX) were assessed as plasma lipid peroxidation biomarkers according to method described by Costa et al, and the advanced oxidation protein products (AOPP) were based on the method described by Witko-Sarsat et al. GSH and GSSG contents were measured using standart kits. Antioxidant enzyme activities, superoxide dismutase (SOD) and catalase (CAT) were determined according to Somani et al and Aebi, respectively.

Cardiovascular functions The evaluation of the participants' cardiovascular responses were made through the Checking of Resting Blood Pressure with the use of a Sphygmomanometer. All measurements were performed with main arm, in triplicate, with patients lying at rest for at least 10 minutes. The heart rate were continuously monitored, after the exercise session, through a cardiac frequency monitor over an hour, every 10 minutes.

Autonomic modulation of the cardiovascular system were analyzed by means of the spectral analysis of heart rate variability. For this, the individuals were in rest, in the pre- and post-exercise moments.

ELIGIBILITY:
Inclusion Criteria:

* Using the Antiretroviral Therapy (ART) for more than six months;
* Have a stabilized clinical picture and viral load.

Exclusion Criteria:

* Physical training programs during the preceding six months;
* Acute or chronic inflammations that could affect the practice of physical exercise;
* Psychiatric disorders;
* Pregnant.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2015-10 (Actual); Primary Completion 2015-12 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
The effect of a short period of supplementation with glutamine dipeptide in the cognitive responses after a resistance training session of women with HIV/AIDS | Before and immediately after a resistance training session
  On the seventh day of supplementation all participants did cognitive function tests before and immediately after a resistance training session.

SECONDARY OUTCOMES:
The effect of a short period of supplementation with glutamine dipeptide in the oxidative stress markers after a resistance training session of women with HIV/AIDS | Before, 1 hour and 2 hours after a resistance training session
  On the seventh day of supplementation all participants had blood collected before, 1 hour and 2 hours after a resistance training session.

CONTACTS AND LOCATIONS:
Overall Officials: Ademar Avelar, PhD, Principal Investigator — University of Maringá

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Somani BL, Ambade V, Bulakh PM, Sharma YV. Elimination of superoxide dismutase interference in fructosamine assay. Clin Biochem. 1999 Apr;32(3):185-8. doi: 10.1016/s0009-9120(99)00016-8. PMID 10383078
- [Background] Aebi H. Catalase in vitro. Methods Enzymol. 1984;105:121-6. doi: 10.1016/s0076-6879(84)05016-3. No abstract available. PMID 6727660
- [Background] Witko-Sarsat V, Friedlander M, Capeillere-Blandin C, Nguyen-Khoa T, Nguyen AT, Zingraff J, Jungers P, Descamps-Latscha B. Advanced oxidation protein products as a novel marker of oxidative stress in uremia. Kidney Int. 1996 May;49(5):1304-13. doi: 10.1038/ki.1996.186. PMID 8731095
- [Background] Nielsen F, Mikkelsen BB, Nielsen JB, Andersen HR, Grandjean P. Plasma malondialdehyde as biomarker for oxidative stress: reference interval and effects of life-style factors. Clin Chem. 1997 Jul;43(7):1209-14. PMID 9216458
- [Derived] de Souza DC, da Silva JC, Matos FO, Okano AH, Bazotte RB, Avelar A. The Effect of a Short Period of Supplementation with Glutamine Dipeptide on the Cognitive Responses after a Resistance Training Session of Women with HIV/AIDS: A Randomized Double-Blind Placebo-Controlled Crossover Study. Biomed Res Int. 2018 Apr 3;2018:2525670. doi: 10.1155/2018/2525670. eCollection 2018. PMID 29850491